CLINICAL TRIAL: NCT05848323
Title: Prospective Case Series to Refine Standalone Cognitive Behavioral Therapy Components for Multiple Sclerosis Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lindsey Knowles, Acting Assistant Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017623
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Multiple sclerosis; Fatigue; Cognitive behavioral therapy; Relaxation training; Behavioral activation; Cognitive therapy
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Relaxation Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relaxation Training (Experimental): Didactic and experiential training in one or more relaxation techniques such as diaphragmatic breathing, progressive muscle relaxation, autogenic relaxation, and guided imagery to reduce autonomic nervous system arousal.
  Interventions: Behavioral: 4-week Relaxation Training
- Behavioral Activation (Experimental): Didactic material and practice focused on identification and reduction of avoidance behaviors (e.g., excessive rest) and increased engagement in valued and reinforcing activities (e.g., physical activity, social engagement).
  Interventions: Behavioral: 4-week Behavioral Activation
- Cognitive Therapy (Experimental): Didactic material and practice focused on identifying, challenging, and modifying inaccurate and/or unhelpful patterns of thought about the self and the world (e.g., catastrophizing the meaning and consequences of fatigue) to change unwanted behavioral patterns (e.g., excessive rest).
  Interventions: Behavioral: 4-week Cognitive Therapy

INTERVENTIONS:
Behavioral: 4-week Relaxation Training — A 4-session telehealth Relaxation Training intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis and the cognitive behavioral model of multiple sclerosis fatigue, b) treatment rationale, b) didactic and experiential training in relaxation techniques such as diaphragmatic breathing, progressive muscle relaxation, autogenic relaxation, and guided imagery, and c) goal setting and problem-solving barriers focused on integrating relaxation practices into daily routine.
  Arms: Relaxation Training
Behavioral: 4-week Behavioral Activation — A 4-session telehealth Behavioral Activation intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis, the cognitive behavioral model of multiple sclerosis fatigue, and self-monitoring activity and energy, b) treatment rationale, c) identification of values/priorities to guide activities, d) activity planning, e) goal setting and problem-solving barriers to engaging in activities.
  Arms: Behavioral Activation
Behavioral: 4-week Cognitive Therapy — A 4-session telehealth Cognitive Therapy intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis, the cognitive behavioral model of multiple sclerosis fatigue, self-monitoring thoughts, and core beliefs, b) treatment rationale, b) labeling thoughts as helpful, unhelpful, or neutral, c) using distraction to cope with unhelpful thoughts, d) challenging and changing unhelpful thoughts, e) problem solving barriers to coping with or changing unhelpful thoughts.
  Arms: Cognitive Therapy

SUMMARY:
This prospective case series will use mixed methods to examine the feasibility, acceptability, and initial effects of three telehealth cognitive behavioral therapy components (relaxation training, behavioral activation, cognitive therapy) for fatigue in people with multiple sclerosis.

DETAILED DESCRIPTION:
Fatigue affects 80% of people with multiple sclerosis (PwMS), and nearly half report fatigue as their most disabling symptom. The cognitive behavioral model of MS fatigue theorizes that MS disease factors trigger fatigue, but fatigue is maintained or worsened by factors like daily stress and how PwMS react cognitively, behaviorally, physiologically, and emotionally to fatigue. In-person and telehealth cognitive behavioral therapy (CBT) for fatigue targets these factors and reactions and is one of the most effective treatments for MS fatigue. However, CBT is resource intensive, as it consists of multiple components (i.e., relaxation training, behavioral activation, cognitive therapy), requiring 8-16 hour-long sessions delivered by a specialized clinician. CBT has yet to be assessed via an integrated translational model that considers all stages, from intervention development to implementation. Thus, the active components of CBT for MS fatigue and their mechanisms are unclear and, despite the significant burden of MS fatigue, CBT for fatigue is not widely accessible due to various implementation barriers.

The proposed prospective case series is the first of two project aims. The overall project aims to optimize CBT for fatigue to maximize efficacy and efficiency. It will use the Multiphase Optimization Strategy to advance scientific evidence on CBT's active components and facilitate implementation, thereby improving accessibility. The proposed prospective case series (Aim 1) will:

1. examine the feasibility and acceptability of telehealth CBT components (relaxation training, behavioral activation, cognitive therapy) for fatigue in PwMS.
2. examine initial effects of telehealth CBT components (relaxation training, behavioral activation, cognitive therapy) for improving fatigue in PwMS.
3. understand participants' perceptions of the feasibility, acceptability, appropriateness, and perceived effectiveness of telehealth CBT components (relaxation training, behavioral activation, cognitive therapy) for improving fatigue in PwMS and their recommendations for improving the CBT components.

ELIGIBILITY:
Inclusion Criteria:

1. MS diagnosis of any subtype per chart review
2. Score 4 or higher on the Fatigue Severity Scale
3. Presence of chronic, problematic fatigue that, in the opinion of the patient, has interfered with their daily activities for 3 or more months
4. Are able to comply with study procedures and complete measures independently assessed via self-report
5. All genders
6. 18 years of age or older
7. Able to read and speak English
8. Are willing to maintain current fatigue treatment regimen for duration of study (although individuals who want to make a change to their fatigue treatment regimen will be considered eligible 3 months after making that change)

Exclusion Criteria:

1. Score greater than 7 on the Patient Determined Disease Steps Scale
2. Has significant cognitive impairment as indicated by 1 or more errors on the 6-item Cognitive Screener
3. Change in disease modifying medications in the prior three months assessed via self-report (although participants will be considered eligible after the 3-month window)
4. History of MS relapse within the last 30 days prior to screening assessed via self-report (although participants will be considered eligible after the 30-day window)
5. Current suicidal ideation with intent or plan as indicated by a score of 1 or higher on the Patient Health Questionnaire-9 suicide item and further assessment with the Columbia-Suicide Severity Rating Scale (although individuals with suicidal ideation but no intent or plan will be considered eligible)
6. Currently engaged in psychotherapy for fatigue assessed via self-report
7. Current pregnancy (although participants will be considered eligible when they are no longer pregnant)
8. Currently participating in another research study that could impact fatigue such as intervention studies targeting mood, energy management, exercise/physical activity, and diet (although participants can be screened for eligibility once they have completed the other research study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Knowles, PhD, Principal Investigator — University of Washington
Locations (1):
- Multiple Sclerosis Center at UW Medical Center - Northwest, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available to interested researchers a data file containing de-identified data used for each published article at the time the article is accepted for publication. The data will be de-identified to remove any variables from which it would be possible to identify any individual participants. Specifically, we will create a data file that includes all variables used in the published article and a list of the variables in the data file (along with variable labels) and send to investigators who request the data a copy of: (1) the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) the dataset (as an SPSS.sav file). Note, though, even though any data files that we share will be stripped of identifiers prior to release for sharing, it remains possible those who access the data could potentially use deduction to identify participants with unusual characteristics or combinations of unusual characteristics.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data used for the analyses for any papers published will become available to interested researchers by request after that article is published. Those data will continue to be available for at least five years following the publication of the article.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a multiple sclerosis comprehensive care center from October 2023 to August 2024.
Pre-assignment Details: Thirty individuals were screened for eligibility. Seven individuals were ineligible due to MS relapse in prior 30 days (n=1), disease modifying therapy change in prior 3 months (n=1), score lower than 4 on the Fatigue Severity Scale (n=3), significant cognitive impairment (n=1), and no MS diagnosis (n=1). One individual declined to participant due to the time commitment for study participation. One individual was excluded because research staff were unable to contact them after several attempts
Period: Overall Study
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Started | 7 | 7 | 7
Completed | 7 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.3) | 47.9 (13.4) | 46.6 (14.9) | 47.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 3 | 2 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 6 | 4 | 3 | 13
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 6 | 6 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Intervention Acceptability
Description: Intervention Acceptability will be measured with the Acceptability of Intervention Measure (AIM). When assessed via online survey, responses from the Intervention Acceptability items are averaged to create a mean score [1-5]. A higher score indicates more agreement with intervention acceptability while a lower score indicates less agreement with intervention acceptability.
Time Frame: Collected via online survey at post-treatment (approximately 4-8 weeks after the pre-treatment survey).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale | 4.36 (0.70) | 4.64 (0.48) | 4.68 (0.59)

2. Primary Outcome: Intervention Appropriateness
Description: Intervention Appropriateness will be measured with the Intervention Appropriateness Measure (IAM). When assessed via online survey, responses from the Intervention Appropriateness items are averaged to create a mean score [1-5]. A higher score indicates more agreement with intervention appropriateness while a lower score indicates less agreement with intervention appropriateness.
Time Frame: Collected via online survey at post-treatment (approximately 4-8 weeks after the pre-treatment survey).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale | 4.14 (0.57) | 4.25 (0.74) | 4.25 (0.78)

3. Primary Outcome: Intervention Feasibility
Description: Intervention Feasibility will be measured with the Feasibility of Intervention Measure (FIM). When assessed via online survey, responses from the Intervention Feasibility items are averaged to create a mean score [1-5]. A higher score indicates more agreement with intervention feasibility while a lower score indicates less agreement with intervention feasibility.
Time Frame: Collected via online survey at post-treatment (approximately 4-8 weeks after the pre-treatment survey).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale | 4.46 (0.57) | 4.39 (0.61) | 4.42 (0.66)

4. Secondary Outcome: Fatigue
Description: Fatigue will be measured by the Modified Fatigue Impact Scale. This is a 21-item self-report questionnaire assessing fatigue-related symptoms in the previous four weeks via 5-point Likert-type scale. It yields a total score (range: 0-84) and a higher score indicates greater fatigue.
Time Frame: Collected via online survey at pre-treatment (up to 4 weeks before treatment session 1) and post-treatment (approximately 4-8 weeks after the pre-treatment survey).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale
  Pre-treatment | 44.29 (11.13) | 49.38 (9.74) | 54.71 (20.15)
  Post-treatment | 36.14 (10.09) | 34.14 (12.27) | 37.29 (13.10)

5. Secondary Outcome: Participation in Social Roles and Activities
Description: Patient Reported Outcomes Measurement Information System Short Form - Ability to Participate in Social Roles and Activities (PROMIS-SRA; Hahn et al., 2010). The 8-item short form version of the PROMIS-SRA assesses the perceived ability to perform one's usual social roles and activities. Items are rated on a 5-point Likert-type scale. Raw summed scores are converted to T-scores standardized to the U.S. general population (mean = 50, standard deviation = 10), with higher scores indicating better ability to participate in social roles and activities.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
T-score
  Pre-treatment | 43.23 (6.09) | 41.39 (5.44) | 40.47 (7.31)
  Post-treatment | 43.64 (4.42) | 46.30 (7.52) | 44.04 (4.28)

6. Secondary Outcome: Relaxation/Serenity
Description: Relaxation/Serenity will be measured by the Positive and Negative Affect Schedule Serenity Subscale. This is a 3-item self-report subscale of the Positive and Negative Affect Schedule assessing perceptions of feeling of calm, relaxed, and at ease over the previous week via a 5-point Likert-type scale. The summed total score ranges from 3-15 and a higher score indicates greater feelings of relaxation/serenity.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale
  Pre-treatment | 9.00 (2.94) | 8.29 (1.38) | 9.57 (4.24)
  Post-treatment | 11.14 (1.95) | 10.00 (2.58) | 11.43 (1.62)

7. Secondary Outcome: Fatigue Catastrophizing
Description: Fatigue catastrophizing will be measured by the Fatigue Catastrophizing Scale. This is a 13-item self-report questionnaire assessing negative beliefs or expectations connected to one's perceptions of fatigue via a 5-point Likert-type scale. Summed total scores range from 0 to 52, and a higher score indicates greater fatigue catastrophizing.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale
  Pre-treatment | 20.57 (9.14) | 18.86 (17.17) | 15.71 (12.79)
  Post-treatment | 19.29 (8.34) | 15.71 (11.25) | 11.43 (7.30)

8. Secondary Outcome: Behavioral Activation
Description: Behavioral activation will be measured by the Behavioral Activation for Depression Scale Short Form. This is a 9-item self-report measure. It assess the extent to which the respondent thinks they have engaged in pleasant and/or goal-directed activity over the past week via a 7-point Likert-type scale. Summed total scores range from 0 to 54, and a higher score indicates greater behavioral activation.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale
  Pre-treatment | 27.14 (4.67) | 24.86 (8.11) | 29.14 (7.34)
  Post-treatment | 27.57 (10.21) | 35.43 (8.02) | 38.43 (6.60)

9. Secondary Outcome: Cognitive Behavioural Responses Questionnaire - Short Form
Description: This is a 18-item self-report questionnaire consisting of five subscales assessing cognitive responses (fear avoidance beliefs, embarrassment avoidance beliefs, symptom focusing) and behavioral responses (resting or avoidance of activity, all-or-nothing behavior) to fatigue one's connected to one's perceptions of fatigue via a 5-point Likert-type scale. The summed total subscale scores range from 0 to 12, and higher scores indicate a more negative response to fatigue.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale
  Fear Avoidance Beliefs at Pre-treatment | 4.00 (2.31) | 5.57 (1.72) | 6.29 (3.55)
  Fear Avoidance Beliefs at Post-treatment | 4.00 (2.08) | 5.57 (1.62) | 4.86 (4.26)
  Embarrassment Avoidance Beliefs at Pre-treatment | 7.57 (3.69) | 6.29 (2.36) | 6.14 (4.06)
  Embarrassment Avoidance Beliefs at Post-treatment | 7.71 (4.39) | 6.14 (4.41) | 6.43 (3.69)
  Symptom Focusing at Pre-treatment | 7.14 (3.34) | 6.43 (2.15) | 6.00 (2.65)
  Symptom Focusing at Post-treatment | 6.57 (3.10) | 4.00 (3.83) | 4.71 (2.21)
  Resting or Avoidance of Activity at Pre-treatment | 4.14 (3.24) | 6.00 (3.16) | 7.29 (3.59)
  Resting or Avoidance of Activity at Post-treatment | 4.14 (3.58) | 5.00 (2.71) | 7.57 (3.26)
  All-or-nothing Behavior at Pre-treatment | 9.00 (2.58) | 10.00 (2.16) | 9.29 (2.29)
  All-or-nothing Behavior at Post-treatment | 8.29 (2.36) | 7.00 (2.38) | 7.43 (3.10)

10. Secondary Outcome: Global Impression of Change
Description: This is a single-item self-report scale that assess the perceived intervention-related change in one's activity limitations, symptoms, emotions, and overall quality of life via 7-point Likert-type scale. The score ranges from 0 to 6 and a higher score indicates greater perceived change.
Time Frame: Collected via online survey at post-treatment (approximately 4-8 weeks after the pre-treatment survey).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
Number analyzed (Participants) | 7 | 7 | 7
Units on a scale | 4.43 (0.98) | 4.29 (1.25) | 4.43 (1.13)

ADVERSE EVENTS:
Time Frame: From enrollment through the treatment period (approximately 4-6 weeks)
Arm/Group | Relaxation Training | Behavioral Activation | Cognitive Therapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT05848323/Prot_000.pdf